CLINICAL TRIAL: NCT00206973
Title: Bronchial Response to Mannitol and Inflammation in Steroid Naive Asthmatics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Other Study IDs: 7654 - man 05
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: mannitol test

SUMMARY:
Study on the relationship between the response of the airways to a bronchial provocation test with mannitol and the degree of airway inflammation in asthma patients.

DETAILED DESCRIPTION:
Study on the relationship between the response of the airways to a bronchial provocation test with mannitol and the degree of airway inflammation in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Steroid naive asthma.
* Non-smoker

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-08; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Celeste porsbjerg, MD, Principal Investigator — unaffilliated
Locations (1):
- Respiratory Research Unit, Med. Clinic I, Bispebjerg Hospital, Bispebjerg Bakke 23, Copenhagen, NV, Denmark